CLINICAL TRIAL: NCT06758258
Title: Evaluating the Impact of Negative Pressure Wound Therapy on Inflammatory Symptom Severity Following Impacted Third Molar Extractions
Brief Title: Negative Pressure Wound Therapy in Oral Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Aras Erdil, Assist. Prof. Dr., Tokat Gaziosmanpasa University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Usak-GOKA-500-500-05
Record Dates: First submitted 2024-12-26; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Edema; Postoperative Pain; Postoperative Complications
Keywords: Negative-Pressure Wound Therapy; Molar, Third
MeSH Terms: conditions — Edema; Pain, Postoperative; Postoperative Complications | interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Intervention Model Description: The study was designed as a randomized controlled parallel-group model. The required sample size will be equally divided into two groups: the study group and the control group. Participants in the study group will receive the targeted therapy, while those in the control group will receive sham appliances under identical conditions.
Who Masked: Participant, Outcomes Assessor
Masking Description: The enrolled participants will be recorded anonymously, with each assigned a unique identification number. These numbers will then be randomized into two study groups using free online randomization software. As a result, both the researcher and the participants will remain blinded to the assigned study groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Negative Pressure Wound Therapy (Experimental): Following third molar extraction, patients receive custom-fit, transparent splints fabricated from thermoformed acrylic resin. Splints are assessed for fit, adaptation, and leak-proof integrity.
  Holes are created in the splints at the surgical site and connected to a physiodispenser irrigation hose using cyanoacrylate adhesive.
  The splint is positioned intraorally, and the physiodispenser pump is operated in reverse to generate negative pressure.
  Personalized negative pressure therapy is applied for three hours, with one-hour sessions
  Interventions: Device: Negative Pressure Wound Therapy
- Sham Therapy (Sham Comparator): All surgical and prosthetic interventions planned for the negative pressure wound therapy (NPWT) arm will be conducted. However, for patients in this arm, while personalized appliances will be placed intraorally, the peristaltic pump of the physiodispenser will remain inactive. The duration (1 hour) and intervals (day of surgery, first and third postoperative days) of appliance application will mirror those of the active NPWT arm.
  Interventions: Device: Sham Therapy

INTERVENTIONS:
Device: Negative Pressure Wound Therapy — Preparations for NPWT:
  1. Impressions & Model:
     Lower jaw impressions were taken with alginate and modified trays for optimal tissue recording.
     Dental plaster models were created.
  2. Splint Fabrication & Connection:
  2mm hard splints were thermoformed and modified for vacuum. Intraoral splint fit was assessed, and soft acrylic ensured an airtight seal. The irrigation hose was connected to the splint via cyanoacrylate adhesive. 3. NPWT Application: The physiodispenser pump was operated in reverse at reduced power (10-20%). Three 1-hour NPWT sessions were performed.
  Arms: Negative Pressure Wound Therapy
Device: Sham Therapy — The same preparations will be conducted for the sham application arm, except that the peristaltic pump of the physiodispenser will remain inactive during application.
  Arms: Sham Therapy

SUMMARY:
Inflammatory complications following the surgical removal of third molars remain a common and unavoidable challenge. These complications significantly impact patients' quality of life, prompting the development of numerous pharmacological and non-pharmacological interventions, as described in the current literature. However, non-interventional and non-pharmacological approaches remain a topic of debate.

Negative pressure wound therapy (NPWT) has demonstrated effectiveness in managing oral cavity wounds, such as orocutaneous and pharyngocutaneous fistulas, as well as drug-induced osteonecrosis. Despite its potential, no clinical studies with a systematic approach have evaluated its use in this context. Therefore, this study aims to assess the effectiveness of NPWT, a method with promising results in wound management, for reducing inflammatory complications following the extraction of impacted third molars, one of the most commonly performed oral surgical procedures.

DETAILED DESCRIPTION:
Impacted tooth surgeries are among the most frequently performed procedures in oral and maxillofacial surgery. These surgeries require intensive training, skill, and experience to minimize trauma during the procedure. Despite careful and atraumatic surgical techniques, complications such as pain, swelling, trismus, and bleeding often occur due to surgical trauma. While these postoperative complications are addressed through atraumatic approaches, their complete elimination remains unattainable. Consequently, numerous studies have been conducted to minimize postoperative inflammatory complications.

According to difficulty level parameters, surgical cases are categorized as uncomplicated, moderately difficult, and difficult. Expected physiological responses to surgical procedures, such as swelling, pain, mild bleeding, and muscle stiffness, may arise depending on these difficulty levels. However, even these expected complications can negatively impact the psychological well-being of patients and cause significant postoperative discomfort.

To alleviate such discomfort and facilitate a smoother recovery, pharmacological treatments, including non-steroidal anti-inflammatory drugs (NSAIDs) and corticosteroids, are commonly administered orally, intramuscularly, or submucosally before or after the procedure. Additionally, extraoral cold applications (e.g., ice packs) are recommended to reduce postoperative edema. However, the effectiveness of ice therapy remains controversial, and no universally accepted non-pharmacological treatment has yet been identified to mitigate expected postoperative inflammatory symptoms.

Negative Pressure Wound Therapy (NPWT) was first introduced in 1986. Its efficacy was demonstrated in an animal study by Morykwas et al. and subsequently in a clinical trial conducted by Argenta and Morykwas in 1997. These promising results led to the development of a systematic device marketed under the name Vacuum Assisted Closure (VAC) by Kinetic Concepts (KCI, San Antonio, TX, USA).

The beneficial effects of NPWT are thought to result from five primary mechanisms: macro tension, micro tension, fluid and edema removal, reduction of infective material, and wound stabilization. Given the inflammatory nature of complications following the surgical extraction of impacted third molars, NPWT is hypothesized to be effective in managing these issues. It is expected that NPWT may accelerate intraoral wound healing, reduce postoperative edema and bacterial load, and consequently improve patients' quality of life after surgery.

To date, there are no observational or interventional studies systematically examining the intraoral application of NPWT. However, some literature suggests its extraoral use in treating orocutaneous and pharyngocutaneous fistulas. Limited case reports have explored intraoral applications, such as in drug-induced jaw necrosis and the decompression of keratocystic lesions, showing promising outcomes.

This study aims to evaluate the effects of NPWT, a non-invasive and non-pharmacological technique, on inflammatory symptoms-pain, swelling, and restricted mouth opening-following the surgical extraction of impacted teeth. Furthermore, instead of employing commercially available NPWT devices, this study seeks to develop and validate a low-cost alternative using readily accessible materials. If successful, this approach could enable broader clinical use of NPWT by dentists and introduce a novel, cost-effective method to the existing literature.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 65 years
* Undergone surgical extraction of a right or left impacted mandibular third molar

Exclusion Criteria:

* Chronic Medical Conditions:

Patients with chronic diseases such as diabetes mellitus, chronic inflammatory diseases, chronic kidney or liver failure, chronic cardiovascular diseases, and autoimmune diseases.

* Immunocompromised Patients:

Immunosuppressed patients, including those diagnosed with malignancy.

* Allergies:

Patients with a history of allergy to any component of the NPWT treatment.

* Non-Adherence:

Patients who did not attend scheduled follow-up appointments within the study protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2024-04-18 (Actual); Primary Completion 2024-10-18 (Actual); Study Completion 2024-11-18 (Actual)

PRIMARY OUTCOMES:
Preoperative Pain Intensity | On the day of surgery preoperatively
  The patients were asked to mark their pain intensities on a Numerical Rating Scale in which '0' means no pain, '5' means moderate pain and '10' means worst imaginable pain on the day of surgery preoperatively.
Change From Baseline Maximal Mouth Opening on Postoperative Follow Up Visits | Preoperatively on the day of surgery, postoperative second and seventh days.
  All patients' maximal mouth opening were measured and recorded as the distance between upper and lower right central incisors.
Change From Baseline Facial Measurements on Postoperative Follow Up Visits | Preoperatively on the day of surgery, postoperative second and seventh days.
  Measurements were performed on the ipsilateral site between tragus and lateral commissura, lateral canthus and angle of mandible with a flexible ruler. The obtained values' average amounts were calculated and recorded for each patient.
Postoperative Pain Intensity-1 | Postoperative Second Day
  The patients were asked to mark their pain intensities on a Numerical Rating Scale in which '0' means no pain, '5' means moderate pain and '10' means worst imaginable pain.
Postoperative Pain Intensity-2 | Postoperative Seventh Day
  The patients were asked to mark their pain intensities on a Numerical Rating Scale in which '0' means no pain, '5' means moderate pain and '10' means worst imaginable pain.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet A Güngör, Prof Dr, Study Chair — Uşak University
Locations (1):
- Tokat Gaziosmanpasa University, Faculty of Dentistry, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Following publication of the study findings in a peer-reviewed journal, requests for data sharing will be considered by the responsible researcher.
Time Frame: Upon publication of the study results
Access Criteria: Reasonable requests

REFERENCES:
- [Background] Sternick M, Gates JC, Champion A, Yampolsky A. Negative pressure wound therapy for complex oral wounds. J Surg Case Rep. 2023 Dec 6;2023(12):rjad638. doi: 10.1093/jscr/rjad638. eCollection 2023 Dec. PMID 38076307
- [Background] Laimer J, Steinmassl O, Hechenberger M, Rasse M, Pikula R, Bruckmoser E. Intraoral Vacuum-Assisted Closure Therapy-A Pilot Study in Medication-Related Osteonecrosis of the Jaw. J Oral Maxillofac Surg. 2017 Oct;75(10):2154-2161. doi: 10.1016/j.joms.2017.02.033. Epub 2017 Mar 18. PMID 28396234
- [Background] Mellott AJ, Zamierowski DS, Andrews BT. Negative Pressure Wound Therapy in Maxillofacial Applications. Dent J (Basel). 2016 Sep 6;4(3):30. doi: 10.3390/dj4030030. PMID 29563472
- [Derived] Erdil A, Celikkol O, Caymaz A, Son A. Effectiveness of topical vacuum assisted drainage in mandibular third molar surgeries: a randomized controlled clinical study. BMC Oral Health. 2025 Nov 25;25(1):1838. doi: 10.1186/s12903-025-07243-0. PMID 41291693